CLINICAL TRIAL: NCT01012245
Title: Project "XCHANGE" Non-Interventional Study
Brief Title: Non-Interventional Study In Patients With Ocular Hypertension And Open Angle Glaucoma Treated With Xalatan And Xalacom
Acronym: XCHANGE
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: 912-OPT-0091-131; A6111100, 912-OPT-0091-131
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2010-01-21 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2010-02

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Xchange; Xalatan; Xalacom; Betablocker; observational; longterm
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with glaucoma and ocular hypertension
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Non-interventional study to obtain real life data from the treatment with Xalatan and Xalacom in Germany and to assess the long-term efficacy and tolerability under routine conditions. Data were entered into an electronic case report form.

ELIGIBILITY:
Inclusion Criteria:

* patients with ocular hypertension or glaucoma, defined by SmPC

Exclusion Criteria:

* defined by SmPC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with glaucoma or ocular hypertension treated by office-based ophthalmologists
Sampling Method: Non-Probability Sample
Enrollment: 28812 (Actual)
Dates: Start 2000-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=912-OPT-0091-131&StudyName=Non-Interventional%20Study%20In%20Patients%20With%20Ocular%20Hypertension%20And%20Open%20Angle%20Glaucoma%20Treated%20With%20Xalatan%20And%20Xalacom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, prospective, multi-center, non-interventional cohort study (NIS) at 385 centers (office-based ophthalmologists); number of subjects per center was not limited.
Pre-assignment Details: Subjects were assigned to a therapeutic strategy within current practice and not according to a protocol.
Groups:
- Subjects With Glaucoma and Ocular Hypertension: All subjects group: documented diagnosis of glaucoma or ocular hypertension at baseline visit; includes subjects from the 4 treatment groups: Xalatan®: subjects with Xalatan® (latanoprost) monotherapy at baseline visit; Betablockers: subjects with only 1 betablocker and subjects with more than one betablocker at baseline visit; Xalacom®: subjects with Xalacom® (latanoprost + timolol maleate) therapy at baseline visit; other medications: subjects with other or no hypotensive therapy at baseline visit.
Period: Overall Study
Arm/Group | Subjects With Glaucoma and Ocular Hypertension
Started | 28812
Completed | 26385 (More than 1 discontinuation (DC) reason possible per subject. See outcome measure Reasons for DC.)
Not Completed | 2427

BASELINE CHARACTERISTICS:
Groups:
- Xalatan®: Subjects with Xalatan® (latanoprost) monotherapy at baseline visit
- Betablockers: Subjects with only 1 betablocker and subjects with more than one betablocker at baseline visit
- Xalacom®: Subjects with Xalacom® (latanoprost + timolol maleate) therapy at baseline visit
- Other Medication: Subjects with other or no hypotensive therapy at baseline visit
- Total: Total of all reporting groups
Arm/Group | Xalatan® | Betablockers | Xalacom® | Other Medication | Total
Number analyzed (Participants) | 13486 | 1884 | 746 | 12696 | 28812
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (13.4) | 65.3 (12.7) | 66.5 (12.7) | 66.9 (13.3) | 65.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7636 | 1101 | 383 | 7493 | 16613
  Male | 5850 | 783 | 363 | 5203 | 12199
Concomitant ocular diseases at baseline [Number; unit: participants] — Number of subjects per type of concomitant ocular diseases present at baseline visit for right eye (OD) and left eye (OS). Column numbers may not equal the total number of participants analyzed as subjects could meet criteria for more than 1 category.
  participants
    Concomitant ocular disease (right eye [OD]) | 13137 | 1846 | 731 | 12328 | 28042
    Concomitant ocular disease (left eye [OS]) | 13179 | 1847 | 732 | 12350 | 28108
    No concomitant diseases OD | 6737 | 1060 | 315 | 4742 | 12854
    No concomitant diseases OS | 6730 | 1067 | 308 | 4757 | 12862
    At least 1 concomitant disease OD | 5426 | 786 | 416 | 6488 | 13116
    At least 1 concomitant disease OS | 5460 | 780 | 424 | 6492 | 13156
    Status post cataract surgery OD | 309 | 39 | 21 | 731 | 1100
    Status post cataract surgery OS | 338 | 40 | 19 | 752 | 1149
    Status post glaucoma surgery OD | 1276 | 189 | 109 | 1799 | 3373
    Status post glaucoma surgery OS | 1292 | 184 | 107 | 1729 | 3312
    Status post laser surgery for glaucoma OD | 656 | 56 | 54 | 1070 | 1836
    Status post laser surgery for glaucoma OS | 637 | 56 | 64 | 1061 | 1818
    Cataract OD | 2297 | 370 | 209 | 2542 | 5418
    Cataract OS | 2302 | 370 | 220 | 2587 | 5479
    Other disease OD | 2249 | 280 | 147 | 2639 | 5315
    Other disease OS | 2269 | 285 | 143 | 2633 | 5330
    Missing values OD | 974 | 0 | 0 | 1098 | 2072
    Missing values OS | 989 | 0 | 0 | 1101 | 2090
Concomitant systemic diseases at baseline [Number; unit: participants] — Number of subjects per type of concomitant systemic disease present at baseline visit. Column numbers may not equal the total number of participants analyzed as subjects could meet criteria for more than one category.
  participants
    No concomitant diseases | 6895 | 1045 | 396 | 5734 | 14070
    At least 1 concomitant disease | 5638 | 839 | 350 | 5854 | 12681
    Diabetes mellitus | 1644 | 247 | 107 | 1743 | 3741
    Asthma | 532 | 43 | 4 | 484 | 1063
    Cardiac insufficiency | 891 | 136 | 48 | 1118 | 2193
    Hypotension | 347 | 75 | 24 | 288 | 734
    Hypertension | 2257 | 453 | 192 | 2288 | 5190
    Other disease | 1696 | 200 | 75 | 1902 | 3873
    Missing values | 953 | 0 | 0 | 1108 | 2061
Glaucoma diagnosis at baseline [Number; unit: participants] — Number of subjects per each type of glaucoma diagnosis present at baseline visit for OD and OS. Column numbers may not equal the total number of participants analyzed as subjects could meet criteria for more than one category.
  participants
    Glaucoma chronicum simplex OD | 9863 | 1595 | 560 | 9266 | 21284
    Glaucoma chronicum simplex OS | 9874 | 1590 | 562 | 9269 | 21295
    Normal tension glaucoma OD | 818 | 51 | 55 | 486 | 1410
    Normal tension glaucoma OS | 834 | 53 | 53 | 507 | 1447
    Chronic narrow-angle glaucoma OD | 496 | 43 | 22 | 804 | 1365
    Chronic narrow-angle glaucoma OS | 503 | 43 | 22 | 804 | 1372
    Congenital glaucoma OD | 26 | 7 | 0 | 58 | 91
    Congenital glaucoma OS | 24 | 8 | 1 | 55 | 88
    Exfoliation glaucoma OD | 339 | 41 | 15 | 381 | 776
    Exfoliation glaucoma OS | 335 | 36 | 16 | 390 | 777
    Pigment dispersion glaucoma OD | 135 | 13 | 8 | 155 | 311
    Pigment dispersion glaucoma OS | 137 | 13 | 9 | 150 | 309
    Neovascular glaucoma OD | 27 | 3 | 5 | 93 | 128
    Neovascular glaucoma OS | 30 | 6 | 5 | 73 | 114
    Other secondary glaucoma OD | 152 | 14 | 18 | 242 | 426
    Other secondary glaucoma OS | 158 | 10 | 16 | 262 | 446
    Acute angle closure OD | 11 | 3 | 0 | 11 | 25
    Acute angle closure OS | 10 | 4 | 0 | 9 | 23
    Ocular hypertension OD | 987 | 60 | 45 | 467 | 1559
    Ocular hypertension OS | 987 | 63 | 46 | 468 | 1564
    Other glaucoma OD | 283 | 16 | 3 | 365 | 667
    Other glaucoma OS | 287 | 21 | 2 | 363 | 673
    No glaucoma OD | 262 | 38 | 14 | 267 | 581
    No glaucoma OS | 230 | 37 | 13 | 259 | 539
    Missing values OD | 87 | 0 | 1 | 101 | 189
    Missing values OS | 77 | 0 | 1 | 87 | 165
Duration of glaucoma disease at baseline [Mean (Standard Deviation); unit: years] — Duration in years for glaucoma disease present at baseline visit.
  years | 5.1 (5.6) | 6.0 (5.9) | 6.6 (6.1) | 6.6 (6.8) | 5.9 (6.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP)
Description: Mean IOP values measured by applanation tonometry. Only Goldman values are displayed; if values were given for both right and left eye, the value of the right eye was analyzed. Change (absolute difference) calculated as mean of (value of IOP at observation minus baseline value). Study course is reported by yearly intervals and clustered as 1 year (12±3 months), 2 years (24±3 months), and 3 years (36±3 months).
Time Frame: Baseline, 1 year, 2 years, and 3 years
Population: All subjects group and each treatment group population. N=number of participants with IOP data at baseline; (n)=number of participants with analyzable data at observation for All subjects, Xalatan®, Betablockers, Xalacom®, and Other medications, respectively.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- All Subjects: Documented diagnosis of glaucoma or ocular hypertension at baseline visit; includes subjects from the 4 treatment groups.
- Other Medications: Subjects with other or no hypotensive therapy at baseline visit.
Arm/Group | All Subjects | Xalatan® | Betablockers | Xalacom® | Other Medications
Number analyzed (Participants) | 20073 | 8735 | 1508 | 494 | 9336
mm Hg
  1 year (n=10886,4134, 357, 209, 3029) | -1.5 (4.4) | -0.7 (3.5) | -1.0 (3.4) | -0.2 (3.5) | -1.1 (4.6)
  2 years (n=7558, 2631, 175, 80, 1834) | -1.6 (4.5) | -0.7 (3.6) | -0.8 (3.2) | -0.5 (3.1) | -1.4 (4.6)
  3 years (n=5023, 1753, 64, 40, 1115) | -1.6 (4.5) | -0.7 (3.7) | -1.2 (3.1) | -0.3 (3.2) | -1.4 (4.4)
Statistical Analysis 1: Comparison: All Subjects; IOP 1 year (n=11602); Test type: Superiority or Other; Mean value = 17.2, 95% CI [17.2 to 17.3], Standard Deviation 3.4
Statistical Analysis 2: Comparison: Xalatan®; IOP 1 year (n=4450); Test type: Superiority or Other; Mean value = 16.9, 95% CI [16.8 to 17.0], Standard Deviation 2.9
Statistical Analysis 3: Comparison: Betablockers; IOP 1 year (n=357); Test type: Superiority or Other; Mean value = 17.3, 95% CI [17.1 to 17.5], Standard Deviation 2.2
Statistical Analysis 4: Comparison: Xalacom®; IOP 1 year (n=220); Test type: Superiority or Other; Mean value = 16.9, 95% CI [16.4 to 17.3], Standard Deviation 3.2
Statistical Analysis 5: Comparison: Other Medications; IOP 1 year (n=3277); Test type: Superiority or Other; Mean value = 17.6, 95% CI [17.5 to 17.8], Standard Deviation 4.1
Statistical Analysis 6: Comparison: All Subjects; IOP 2 years (n=8051); Test type: Superiority or Other; Mean value = 17.0, 95% CI [17.0 to 17.1], Standard Deviation 3.4
Statistical Analysis 7: Comparison: Xalatan®; IOP 2 years (n=2808); Test type: Superiority or Other; Mean value = 16.8, 95% CI [16.7 to 16.9], Standard Deviation 2.9
Statistical Analysis 8: Comparison: Betablockers; IOP 2 years (n=175); Test type: Superiority or Other; Mean value = 17.2, 95% CI [17.0 to 17.5], Standard Deviation 1.8
Statistical Analysis 9: Comparison: Xalacom®; IOP 2 years (n=83); Test type: Superiority or Other; Mean value = 16.6, 95% CI [15.9 to 17.2], Standard Deviation 2.8
Statistical Analysis 10: Comparison: Other Medications; IOP 2 years (n=2002); Test type: Superiority or Other; Mean value = 17.1, 95% CI [16.9 to 17.2], Standard Deviation 3.7
Statistical Analysis 11: Comparison: All Subjects; IOP 3 years (n=5469); Test type: Superiority or Other; Mean value = 17.0, 95% CI [16.9 to 17.1], Standard Deviation 3.4
Statistical Analysis 12: Comparison: Xalatan®; IOP 3 years (n=1932); Test type: Superiority or Other; Mean value = 16.8, 95% CI [16.7 to 17.0], Standard Deviation 3.2
Statistical Analysis 13: Comparison: Betablockers; IOP 3 years (n=64); Test type: Superiority or Other; Mean value = 17.5, 95% CI [16.9 to 18.1], Standard Deviation 2.5
Statistical Analysis 14: Comparison: Xalacom®; IOP 3 years (n=44); Test type: Superiority or Other; Mean value = 16.5, 95% CI [15.7 to 17.4], Standard Deviation 2.8
Statistical Analysis 15: Comparison: Other Medications; IOP 3 years (n=1251); Test type: Superiority or Other; Mean value = 16.9, 95% CI [16.7 to 17.1], Standard Deviation 3.6

2. Primary Outcome: Aulhorn Stage (Visual Field Defects)
Description: Number of subjects at each Aulhorn stage. Staged as: No scotoma; Stage I (relative scotomas only), Stage II (absolute scotomas without connection to the blind spot), Stage III (absolute scotomas with connection to the blind spot), Stage IV (absolute scotomas more than 1 quadrant affected), and Stage V (temporal residual visual field only). If values were given for both right and left eye, the value of the right eye was analyzed.
Time Frame: Baseline, 1 year, 2 years, and 3 years
Population: All subjects group and all treatment groups populations
Measure: Number; unit: participants
Arm/Group | All Subjects | Xalatan® | Betablockers | Xalacom® | Other Medications
Number analyzed (Participants) | 28812 | 13486 | 1884 | 746 | 12696
participants
  Baseline: No scotoma | 7753 | 4074 | 493 | 200 | 2986
  Baseline: Stage I | 3759 | 1915 | 254 | 68 | 1522
  Baseline: Stage II | 1904 | 826 | 119 | 47 | 912
  Baseline: Stage III | 1313 | 467 | 51 | 57 | 738
  Baseline: Stage IV | 949 | 268 | 29 | 17 | 635
  Baseline: Stage V | 646 | 210 | 13 | 8 | 415
  Baseline: missing values | 12488 | 5726 | 925 | 349 | 5488
  1 year: No scotoma | 4493 | 2068 | 157 | 94 | 903
  1 year: Stage I | 1763 | 840 | 24 | 23 | 423
  1 year: Stage II | 868 | 326 | 9 | 18 | 279
  1 year: Stage III | 576 | 180 | 3 | 12 | 259
  1 year: Stage IV | 372 | 83 | 1 | 9 | 204
  1 year: Stage V | 212 | 57 | 1 | 3 | 112
  1 year: missing values | 8820 | 3438 | 171 | 168 | 2342
  2 years: No scotoma | 3374 | 1491 | 121 | 43 | 572
  2 years: Stage I | 1339 | 583 | 13 | 8 | 287
  2 years: Stage II | 603 | 193 | 3 | 7 | 190
  2 years: Stage III | 396 | 120 | 0 | 4 | 162
  2 years: Stage IV | 241 | 53 | 1 | 0 | 124
  2 years: Stage V | 141 | 34 | 2 | 1 | 61
  2 years: missing values | 6107 | 2181 | 40 | 76 | 1471
  3 years: No scotoma | 2323 | 1017 | 16 | 21 | 347
  3 years: Stage I | 933 | 416 | 10 | 5 | 185
  3 years: Stage II | 420 | 132 | 7 | 2 | 120
  3 years: Stage III | 288 | 82 | 3 | 1 | 119
  3 years: Stage IV | 173 | 38 | 2 | 2 | 89
  3 years: Stage V | 80 | 17 | 0 | 0 | 35
  3 years: missing values | 4283 | 1515 | 26 | 32 | 924

3. Primary Outcome: Change From Baseline in Optic Disc Excavation: Vertical Cup to Disc Ratio
Description: Mean vertical cup to disc (cup/disc or C/D) ratio to assess the progression of glaucoma; calculated as the ratio of the diameter of the depression (cup) to that of the optical nerve head (disc). If values were given for both right and left eye, the value of the right eye was analyzed. Change calculated as mean of (value of cup/disc ratio at observation minus baseline value).
Time Frame: Baseline, 1 year, 2 years, and 3 years
Population: All subjects group and all treatment groups populations. N=number of participants with optic disc excavation data at baseline; (n)=number of participants with analyzable data at observation for All subjects, Xalatan®, Betablockers, Xalacom®, and Other medications, respectively.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Subjects | Xalatan® | Betablockers | Xalacom® | Other Medications
Number analyzed (Participants) | 20375 | 9521 | 1276 | 497 | 9081
ratio
  1 year (n=11190, 4638, 72, 236, 2714) | 0.00 (0.07) | 0.00 (0.07) | 0.02 (0.08) | 0.01 (0.07) | 0.00 (0.08)
  2 years (n=8088, 3128, 26, 93, 1756) | 0.01 (0.08) | 0.01 (0.08) | 0.00 (0.09) | 0.02 (0.07) | 0.01 (0.08)
  3 years (n=5784, 2173, 16, 34, 1170) | 0.01 (0.09) | 0.01 (0.08) | 0.03 (0.09) | 0.02 (0.11) | 0.01 (0.10)
Statistical Analysis 1: Comparison: All Subjects; Vertical C/D ratio 1 year (n=11966); Test type: Superiority or Other; Mean value = 0.46, 95% CI [0.46 to 0.47], Standard Deviation 0.25
Statistical Analysis 2: Comparison: Xalatan®; Vertical C/D ratio 1 year (n=4944); Test type: Superiority or Other; Mean value = 0.44, 95% CI [0.43 to 0.44], Standard Deviation 0.24
Statistical Analysis 3: Comparison: Betablockers; Vertical C/D ratio 1 year (n=88); Test type: Superiority or Other; Mean value = 0.39, 95% CI [0.35 to 0.43], Standard Deviation 0.19
Statistical Analysis 4: Comparison: Xalacom®; Vertical C/D ratio 1 year (n=241); Test type: Superiority or Other; Mean value = 0.50, 95% CI [0.47 to 0.53], Standard Deviation 0.24
Statistical Analysis 5: Comparison: Other Medications; Vertical C/D ratio 1 year (n=2949); Test type: Superiority or Other; Mean value = 0.51, 95% CI [0.50 to 0.52], Standard Deviation 0.27
Statistical Analysis 6: Comparison: All Subjects; Vertical C/D ratio 2 years (n=8783); Test type: Superiority or Other; Mean value = 0.46, 95% CI [0.46 to 0.47], Standard Deviation 0.25
Statistical Analysis 7: Comparison: Xalatan®; Vertical C/D ratio 2 years (n=3396); Test type: Superiority or Other; Mean value = 0.43, 95% CI [0.42 to 0.44], Standard Deviation 0.23
Statistical Analysis 8: Comparison: Betablockers; Vertical C/D ratio 2 years (n=31); Test type: Superiority or Other; Mean value = 0.39, 95% CI [0.33 to 0.45], Standard Deviation 0.16
Statistical Analysis 9: Comparison: Xalacom®; Vertical C/D ratio 2 years (n=95); Test type: Superiority or Other; Mean value = 0.49, 95% CI [0.44 to 0.54], Standard Deviation 0.24
Statistical Analysis 10: Comparison: Other Medications; Vertical C/D ratio 2 years (n=1934); Test type: Superiority or Other; Mean value = 0.51, 95% CI [0.50 to 0.53], Standard Deviation 0.27
Statistical Analysis 11: Comparison: All Subjects; Vertical C/D ratio 3 years (n=6344); Test type: Superiority or Other; Mean value = 0.45, 95% CI [0.44 to 0.45], Standard Deviation 0.24
Statistical Analysis 12: Comparison: Xalatan®; Vertical C/D ratio 3 years (n=2372); Test type: Superiority or Other; Mean value = 0.42, 95% CI [0.41 to 0.43], Standard Deviation 0.22
Statistical Analysis 13: Comparison: Betablockers; Vertical C/D ratio 3 years (n=25); Test type: Superiority or Other; Mean value = 0.33, 95% CI [0.27 to 0.39], Standard Deviation 0.14
Statistical Analysis 14: Comparison: Xalacom®; Vertical C/D ratio 3 years (n=36); Test type: Superiority or Other; Mean value = 0.47, 95% CI [0.41 to 0.53], Standard Deviation 0.18
Statistical Analysis 15: Comparison: Other Medications; Vertical C/D ratio 3 years (n=1283); Test type: Superiority or Other; Mean value = 0.49, 95% CI [0.48 to 0.51], Standard Deviation 0.26

4. Primary Outcome: Change From Baseline in Optic Disc Excavation: Horizontal Cup to Disc Ratio
Description: Mean horizontal cup to disc (cup/disc or C/D) ratio to assess the progression of glaucoma; calculated as the ratio of the diameter of the depression (cup) to that of the optical nerve head (disc). If values were given for both right and left eye, the value of the right eye was analyzed. Change calculated as mean of (value of cup/disc ratio at observation minus baseline value).
Time Frame: Baseline, 1 year, 2 years, and 3 years
Population: All subjects group and all treatment groups populations. N=number of subjects with optic disc excavation data at baseline; (n)=number of subjects with analyzable data at observation for All subjects, Xalatan®, Betablockers, Xalacom®, and Other medications, respectively.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Subjects | Xalatan® | Betablockers | Xalacom® | Other Medications
Number analyzed (Participants) | 19316 | 9203 | 1226 | 469 | 8418
ratio
  1 year (n=10602, 4496, 71, 227, 2442) | 0.00 (0.07) | 0.00 (0.06) | 0.02 (0.08) | 0.01 (0.07) | 0.00 (0.08)
  2 years (n=7727, 3003, 26, 88, 1630) | 0.00 (0.08) | 0.00 (0.07) | 0.00 (0.10) | 0.01 (0.06) | 0.01 (0.09)
  3 years (n=5500, 2089, 16, 33, 1067) | 0.01 (0.09) | 0.01 (0.07) | 0.01 (0.08) | 0.02 (0.11) | 0.01 (0.10)
Statistical Analysis 1: Comparison: All Subjects; Horizontal C/D ratio 1 year (n=11433); Test type: Superiority or Other; Mean value = 0.45, 95% CI [0.45 to 0.46], Standard Deviation 0.25
Statistical Analysis 2: Comparison: Xalatan®; Horizontal C/D ratio 1 year (n=4810); Test type: Superiority or Other; Mean value = 0.42, 95% CI [0.42 to 0.43], Standard Deviation 0.23
Statistical Analysis 3: Comparison: Betablockers; Horizontal C/D ratio 1 year (n=87); Test type: Superiority or Other; Mean value = 0.37, 95% CI [0.33 to 0.42], Standard Deviation 0.19
Statistical Analysis 4: Comparison: Xalacom®; Horizontal C/D ratio 1 year (n=232); Test type: Superiority or Other; Mean value = 0.50, 95% CI [0.47 to 0.53], Standard Deviation 0.25
Statistical Analysis 5: Comparison: Other Medications; Horizontal C/D ratio 1 year (n=2703); Test type: Superiority or Other; Mean value = 0.51, 95% CI [0.50 to 0.52], Standard Deviation 0.27
Statistical Analysis 6: Comparison: All Subjects; Horizontal C/D ratio 2 years (n=8427); Test type: Superiority or Other; Mean value = 0.45, 95% CI [0.44 to 0.45], Standard Deviation 0.25
Statistical Analysis 7: Comparison: Xalatan®; Horizontal C/D ratio 2 years (n=3276); Test type: Superiority or Other; Mean value = 0.41, 95% CI [0.40 to 0.42], Standard Deviation 0.23
Statistical Analysis 8: Comparison: Betablockers; Horizontal C/D ratio 2 years (n=31); Test type: Superiority or Other; Mean value = 0.38, 95% CI [0.31 to 0.45], Standard Deviation 0.19
Statistical Analysis 9: Comparison: Xalacom®; Horizontal C/D ratio 2 years (n=92); Test type: Superiority or Other; Mean value = 0.50, 95% CI [0.45 to 0.56], Standard Deviation 0.25
Statistical Analysis 10: Comparison: Other Medications; Horizontal C/D ratio 2 years (n=1812); Test type: Superiority or Other; Mean value = 0.51, 95% CI [0.49 to 0.52], Standard Deviation 0.27
Statistical Analysis 11: Comparison: All Subjects; Horizontal C/D ratio 3 years (n=6102); Test type: Superiority or Other; Mean value = 0.43, 95% CI [0.43 to 0.44], Standard Deviation 0.24
Statistical Analysis 12: Comparison: Xalatan®; Horizontal C/D ratio 3 years (n=2289); Test type: Superiority or Other; Mean value = 0.40, 95% CI [0.39 to 0.41], Standard Deviation 0.22
Statistical Analysis 13: Comparison: Betablockers; Horizontal C/D ratio 3 years (n=25); Test type: Superiority or Other; Mean value = 0.31, 95% CI [0.25 to 0.38], Standard Deviation 0.15
Statistical Analysis 14: Comparison: Xalacom®; Horizontal C/D ratio 3 years (n=35); Test type: Superiority or Other; Mean value = 0.49, 95% CI [0.42 to 0.57], Standard Deviation 0.21
Statistical Analysis 15: Comparison: Other Medications; Horizontal C/D ratio 3 years (n=1204); Test type: Superiority or Other; Mean value = 0.48, 95% CI [0.47 to 0.50], Standard Deviation 0.26

5. Secondary Outcome: Investigator Assessment of Xalatan® Efficacy
Description: Number of subjects for Investigator assessment of the efficacy of Xalatan® treatment rated as excellent (highly effective), very good, good, moderate, sufficient, and insufficient (not effective).
Time Frame: Baseline, 1 year, 2 years, and 3 years
Population: Xalatan® treatment group only (subjects with Xalatan® monotherapy at baseline visit).
Measure: Number; unit: participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 13486
participants
  Baseline: Excellent | 555
  Baseline: Very good | 978
  Baseline: Good | 538
  Baseline: Moderate | 92
  Baseline: Sufficient | 15
  Baseline: Insufficient | 23
  Baseline: missing values | 11285
  1 year: Excellent | 910
  1 year: Very good | 3216
  1 year: Good | 2489
  1 year: Moderate | 310
  1 year: Sufficient | 30
  1 year: Insufficient | 34
  1 year: missing values | 3
  2 years: Excellent | 475
  2 years: Very good | 2153
  2 years: Good | 1828
  2 years: Moderate | 164
  2 years: Sufficient | 23
  2 years: Insufficient | 10
  2 years: missing values | 2
  3 years: Excellent | 256
  3 years: Very good | 1548
  3 years: Good | 1307
  3 years: Moderate | 74
  3 years: Sufficient | 19
  3 years: Insufficient | 11
  3 years: missing values | 2

6. Secondary Outcome: Subject Assessment of Satisfaction With Xalatan® Treatment
Description: Number of subjects for assessment of subject satisfaction with Xalatan® treatment; categorized as excellent (full satisfaction), very good, good, moderate, sufficient, and insufficient (no satisfaction).
Time Frame: Baseline, 1 year, 2 years, and 3 years
Population: Xalatan® treatment group only (subjects with Xalatan monotherapy at baseline visit).
Measure: Number; unit: participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 13486
participants
  Baseline: Excellent | 901
  Baseline: Very good | 737
  Baseline: Good | 404
  Baseline: Moderate | 35
  Baseline: Sufficient | 110
  Baseline: Insufficient | 7
  Baseline: missing values | 11292
  1 year: Excellent | 1078
  1 year: Very good | 3200
  1 year: Good | 2510
  1 year: Moderate | 169
  1 year: Sufficient | 16
  1 year: Insufficient | 16
  1 year: missing values | 3
  2 years: Excellent | 621
  2 years: Very good | 2082
  2 years: Good | 1832
  2 years: Moderate | 106
  2 years: Sufficient | 8
  2 years: Insufficient | 4
  2 years: missing values | 2
  3 years: Excellent | 343
  3 years: Very good | 1499
  3 years: Good | 1309
  3 years: Moderate | 54
  3 years: Sufficient | 7
  3 years: Insufficient | 3
  3 years: missing values | 2

7. Secondary Outcome: Visual Acuity (Visus)
Description: Number of subjects with visual acuity evaluations: amaurosis (partial or total loss of sight); hand movements (able to detect gross object and motion perception without detailed discrimination); finger count (able to count fingers at a given distance); visual acuity scale: range 0.05 (low acuity) to >1.2 (greater acuity). If values were given for both the right eye and left eye, the value of the right eye was analyzed.
Time Frame: Baseline, 1 year, 2 years, and 3 years
Population: All subjects group and all treatment groups populations
Measure: Number; unit: participants
Arm/Group | All Subjects | Xalatan® | Betablockers | Xalacom® | Other Medications
Number analyzed (Participants) | 28812 | 13486 | 1884 | 746 | 12696
participants
  Baseline: Amaurosis | 16 | 4 | 1 | 1 | 10
  Baseline: Hand movements | 503 | 176 | 28 | 15 | 284
  Baseline: Finger count | 241 | 94 | 15 | 9 | 123
  Baseline: 0.05 | 766 | 238 | 17 | 26 | 485
  Baseline: 0.1 | 553 | 194 | 25 | 11 | 323
  Baseline: 0.2 | 759 | 308 | 40 | 12 | 399
  Baseline: 0.3 | 902 | 355 | 50 | 27 | 470
  Baseline: 0.4 | 1345 | 567 | 62 | 33 | 683
  Baseline: 0.5 | 2173 | 941 | 138 | 56 | 1038
  Baseline: 0.6 | 2780 | 1242 | 217 | 84 | 1237
  Baseline: 0.7 | 1799 | 846 | 107 | 41 | 805
  Baseline: 0.8 | 4984 | 2329 | 395 | 132 | 2128
  Baseline: 0.9 | 1880 | 928 | 130 | 50 | 772
  Baseline: 1.0 | 8685 | 4505 | 613 | 222 | 3345
  Baseline: 1.1 | 62 | 42 | 8 | 1 | 11
  Baseline: 1.2 | 513 | 258 | 23 | 13 | 219
  Baseline: >1.2 | 117 | 77 | 1 | 5 | 34
  Baseline: Missing values | 734 | 382 | 14 | 8 | 330
  1 year: Amaurosis | 9 | 0 | 0 | 1 | 4
  1 year: Hand movements | 319 | 97 | 1 | 5 | 153
  1 year: Finger counts | 179 | 51 | 5 | 6 | 79
  1 year: 0.05 | 291 | 86 | 2 | 9 | 120
  1 year: 0.1 | 238 | 74 | 3 | 7 | 79
  1 year: 0.2 | 381 | 127 | 9 | 4 | 146
  1 year: 0.3 | 484 | 160 | 9 | 7 | 180
  1 year: 0.4 | 720 | 270 | 7 | 13 | 233
  1 year: 0.5 | 1225 | 463 | 19 | 23 | 334
  1 year: 0.6 | 1663 | 625 | 68 | 38 | 494
  1 year: 0.7 | 1087 | 418 | 1 | 23 | 301
  1 year: 0.8 | 2872 | 1161 | 116 | 57 | 697
  1 year: 0.9 | 1152 | 489 | 5 | 26 | 224
  1 year: 1.0 | 4687 | 2242 | 106 | 78 | 844
  1 year: 1.1 | 39 | 28 | 0 | 0 | 4
  1 year: 1.2 | 322 | 152 | 0 | 5 | 70
  1 year: >1.2 | 52 | 28 | 1 | 2 | 5
  1 year: Missing values | 1384 | 521 | 14 | 23 | 555
  2 years: Amaurosis | 9 | 1 | 0 | 1 | 0
  2 years: Hand movements | 214 | 53 | 0 | 2 | 87
  2 years: Finger counts | 126 | 31 | 4 | 1 | 49
  2 years: 0.05 | 191 | 41 | 0 | 4 | 80
  2 years: 0.1 | 188 | 52 | 0 | 3 | 71
  2 years: 0.2 | 263 | 72 | 4 | 2 | 90
  2 years: 0.3 | 351 | 111 | 0 | 3 | 108
  2 years: 0.4 | 470 | 150 | 3 | 6 | 145
  2 years: 0.5 | 856 | 309 | 5 | 14 | 210
  2 years: 0.6 | 1167 | 385 | 41 | 16 | 327
  2 years: 0.7 | 738 | 255 | 2 | 5 | 162
  2 years: 0.8 | 2051 | 775 | 63 | 28 | 424
  2 years: 0.9 | 900 | 352 | 4 | 9 | 160
  2 years 1.0 | 3437 | 1607 | 50 | 33 | 536
  2 years: 1.1 | 29 | 22 | 0 | 0 | 1
  2 years: 1.2 | 234 | 97 | 0 | 4 | 41
  2 years: >1.2 | 22 | 7 | 0 | 1 | 3
  2 years: Missing values | 955 | 335 | 4 | 7 | 373
  3 years: Amaurosis | 4 | 1 | 0 | 0 | 2
  3 years: Hand movements | 133 | 33 | 2 | 0 | 47
  3 years: Finger counts | 82 | 26 | 0 | 0 | 26
  3 years: 0.05 | 134 | 26 | 0 | 2 | 57
  3 years: 0.1 | 137 | 34 | 3 | 3 | 43
  3 years: 0.2 | 194 | 53 | 1 | 1 | 61
  3 years: 0.3 | 227 | 65 | 4 | 0 | 74
  3 years: 0.4 | 342 | 107 | 3 | 5 | 89
  3 years: 0.5 | 606 | 207 | 8 | 5 | 136
  3 years: 0.6 | 789 | 258 | 7 | 9 | 190
  3 years: 0.7 | 534 | 185 | 3 | 1 | 111
  3 years: 0.8 | 1369 | 538 | 16 | 19 | 260
  3 years: 0.9 | 593 | 210 | 1 | 3 | 85
  3 years: 1.0 | 2487 | 1147 | 16 | 13 | 347
  3 years: 1.1 | 24 | 18 | 0 | 0 | 1
  3 years: 1.2 | 170 | 61 | 0 | 1 | 32
  3 years: >1.2 | 13 | 5 | 0 | 1 | 0
  3 years: Missing values | 662 | 243 | 0 | 0 | 258

8. Secondary Outcome: Visual Impairment Due to Glaucoma
Description: Number of subjects per level of visual impairment categorized as not at all (no impairment), a little bit, moderate, severe, and very severe (very severe impairment).
Time Frame: Baseline, 1 year, 2 years, and 3 years
Population: All subjects group; not summarized by subgroups
Measure: Number; unit: participants
Groups:
- All Subjects: Documented diagnosis of glaucoma or ocular hypertension and a documented glaucoma medication at baseline visit.
Arm/Group | All Subjects
Number analyzed (Participants) | 28812
participants
  Baseline: Not at all | 9368
  Baseline: A little bit | 5171
  Baseline: Moderate | 1723
  Baseline: Severe | 627
  Baseline: Very severe | 235
  Baseline: Missing values | 11688
  1 year: Not at all | 7184
  1 year: A little bit | 4269
  1 year: Moderate | 836
  1 year: Severe | 284
  1 year: Very severe | 91
  1 year: Missing values | 4440
  2 years: Not at all | 4917
  2 years: A little bit | 2961
  2 years: Moderate | 715
  2 years: Severe | 156
  2 years: Very severe | 50
  2 years: Missing values | 3402
  3 years: Not at all | 3120
  3 years: A little bit | 2137
  3 years: Moderate | 501
  3 years: Severe | 110
  3 years: Very severe | 48
  3 years: Missing values | 2584

9. Secondary Outcome: Subject Self-care: Application of Eye Drops
Description: Number of subjects per level of ability for application (administration) of eye drops categorized as without the help of nursing staff (apply without help) and with the help of nursing staff (apply with help).
Time Frame: Baseline, 1 year, 2 years, and 3 years
Population: All subjects group; not summarized by subgroups
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 28812
participants
  Baseline: apply without help | 16520
  Baseline: apply with help | 1142
  Baseline: missing values | 11150
  1 year: apply without help | 12415
  1 year: apply with help | 919
  1 year: missing values | 3770
  2 years: apply without help | 8657
  2 years: apply with help | 391
  2 years: missing values | 3153
  3 years: apply without help | 5829
  3 years: apply with help | 265
  3 years: missing values | 2406

10. Secondary Outcome: Reasons for Changes in Glaucoma Therapy
Description: Number of subjects for each reason for change of therapy; there may be more than one reason possible per patient. Reasons for changes in glaucoma therapy was reported from January 2000 through December 2008 independent of the duration of any individual subject's time on study.
Time Frame: January 2000 through December 2008
Population: Subjects from the all subjects group that changed therapy through the duration of the study; subjects who changed from or changed to "other" therapy (Other Medication) were not included in this analysis; not summarized by subgroups.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 8895
participants
  Wish for better compliance | 1055
  Wish for stronger IOP decrease | 3474
  Wish for better local tolerability | 787
  Wish for better systemic tolerability | 504
  No medication until now | 490
  Other reason | 284
  Missing values | 3859

11. Secondary Outcome: Investigator Assessment of Tolerability of Xalatan® Treatment
Description: Number of subjects for the Investigator's assessment of subjects tolerability of Xalatan® treatment categorized as excellent, very good, good, moderate, sufficient, or insufficient. The occurrence of adverse events (a side effect that may not have any causal relationship to study treatment) was documented as tolerability data.
Time Frame: Baseline up to 3 years
Population: Xalatan® treatment group only (subjects with Xalatan monotherapy at baseline visit).
Measure: Number; unit: participants
Arm/Group | Xalatan®
Number analyzed (Participants) | 13486
participants
  Baseline: Excellent | 619
  Baseline: Very good | 1075
  Baseline: Good | 449
  Baseline: Moderate | 45
  Baseline: Sufficient | 4
  Baseline: Insufficient | 9
  Baseline: Missing values | 11285
  1 year: Excellent | 986
  1 year: Very good | 3429
  1 year: Good | 2437
  1 year: Moderate | 110
  1 year: Sufficient | 18
  1 year: Insufficient | 9
  1 year: Missing values | 3
  2 years: Excellent | 550
  2 years: Very good | 2203
  2 years: Good | 1795
  2 years: Moderate | 96
  2 years: Sufficient | 7
  2 years: Insufficient | 2
  2 years: Missing values | 2
  3 years: Excellent | 284
  3 years: Very good | 1571
  3 years: Good | 1281
  3 years: Moderate | 69
  3 years: Sufficient | 8
  3 years: Insufficient | 2
  3 years: Missing values | 2

12. Secondary Outcome: Reasons for Discontinuation From Study
Description: Number of subjects per reason for discontinuation from the study. More than one reason for discontinuation is possible per patient. Discontinuation analysis was performed independent of the duration of any individual subject's time on study.
Time Frame: January 2000 through December 2008
Population: Subjects from the All subjects group population who discontinued the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 2427
participants
  Lost to follow-up | 717
  Subject's death | 589
  Subject moved | 320
  Adverse event | 337
  Other reason | 302

13. Secondary Outcome: Changes to the Color of the Iris During Xalatan® or Xalacom® Treatment
Description: Number of subjects with documented change to the color of the iris during treatment with Xalatan® or Xalacom®.
Time Frame: Baseline up to 3 years
Population: Xalatan® treatment group (subjects with Xalatan® (latanoprost) monotherapy at baseline visit) and Xalacom® treatment group (latanoprost + timolol maleate) therapy at baseline visit. During the course of the study the data structure (scaling of color) was changed in a way that change in iris color was no longer evaluable; data not summarized.
Arm/Group | Xalatan® | Xalacom®
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data for Adverse drug reactions was reported January 2000 through December 2008 through the duration of the study independent of the duration of any individual subject's time on study.
Description: Side effects = Adverse drug reactions: determination by the health-care professional of causal relationship between occurrence of side effect and drug being used; includes ocular and systemic side effects. Reported for All subjects group population.
Groups:
- All Subjects: Subjects with documented diagnosis of glaucoma or ocular hypertension at baseline visit.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/28812
Other Adverse Events (participants affected / at risk) | 6936/28812
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=28812)
Angina pectoris (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 220
Bradycardia (Cardiac disorders) | 9
Cardiac discomfort (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 9
Cyanosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Anophthalmos (Congenital, familial and genetic disorders) | 6
Developmental glaucoma (Congenital, familial and genetic disorders) | 1
Distichiasis (Congenital, familial and genetic disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Vertigo (Ear and labyrinth disorders) | 6
Goitre (Endocrine disorders) | 2
Abnormal sensation in eye (Eye disorders) | 12
Accommodation disorder (Eye disorders) | 1
Acquired corneal dystrophy (Eye disorders) | 1
Amblyopia (Eye disorders) | 2
Angle closure glaucoma (Eye disorders) | 1
Anterior capsule contraction (Eye disorders) | 1
Anterior chamber disorder (Eye disorders) | 1
Asthenopia (Eye disorders) | 4
Astigmatism (Eye disorders) | 1
Blepharitis (Eye disorders) | 15
Cataract (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 2
Conjunctival hyperaemia (Eye disorders) | 4
Conjunctival irritation (Eye disorders) | 7
Conjunctival oedema (Eye disorders) | 1
Conjunctival pigmentation (Eye disorders) | 2
Conjunctivitis (Eye disorders) | 4
Corneal decompensation (Eye disorders) | 1
Corneal defect (Eye disorders) | 1
Corneal disorder (Eye disorders) | 1
Corneal epithelium defect (Eye disorders) | 3
Corneal erosion (Eye disorders) | 4
Corneal hypertrophy (Eye disorders) | 1
Corneal infiltrates (Eye disorders) | 2
Corneal oedema (Eye disorders) | 5
Corneal opacity (Eye disorders) | 1
Corneal pigmentation (Eye disorders) | 1
Corneal thinning (Eye disorders) | 5
Cyanopsia (Eye disorders) | 1
Dark circles under eyes (Eye disorders) | 2
Diplopia (Eye disorders) | 2
Dry eye (Eye disorders) | 16
Ectropion (Eye disorders) | 1
Eczema eyelids (Eye disorders) | 5
Entropion (Eye disorders) | 1
Erythema of eyelid (Eye disorders) | 14
Eye discharge (Eye disorders) | 7
Eye inflammation (Eye disorders) | 1
Eye irritation (Eye disorders) | 2252
Eye oedema (Eye disorders) | 1
Eye pain (Eye disorders) | 17
Eye pruritus (Eye disorders) | 31
Eye swelling (Eye disorders) | 1
Eyelash discolouration (Eye disorders) | 10
Eyelid oedema (Eye disorders) | 7
Eyelid ptosis (Eye disorders) | 1
Eyelid sensory disorder (Eye disorders) | 2
Eyelids pruritus (Eye disorders) | 3
Foreign body sensation in eyes (Eye disorders) | 1150
Growth of eyelashes (Eye disorders) | 148
Hypermetropia (Eye disorders) | 1
Hyphaema (Eye disorders) | 1
Hypoaesthesia eye (Eye disorders) | 2
Iris disorder (Eye disorders) | 1
Iris hyperpigmentation (Eye disorders) | 21
Iris hypopigmentation (Eye disorders) | 1
Iritis (Eye disorders) | 1
Keratitis (Eye disorders) | 4
Keratoconjunctivitis sicca (Eye disorders) | 4
Lacrimation increased (Eye disorders) | 50
Macular degeneration (Eye disorders) | 2
Macular oedema (Eye disorders) | 9
Maculopathy (Eye disorders) | 3
Miosis (Eye disorders) | 56
Mydriasis (Eye disorders) | 1
Myodesopsia (Eye disorders) | 2
Myopia (Eye disorders) | 1
Night blindness (Eye disorders) | 2
Ocular hyperaemia (Eye disorders) | 3760
Optic disc haemorrhage (Eye disorders) | 1
Optic nerve cupping (Eye disorders) | 1
Photophobia (Eye disorders) | 5
Photopsia (Eye disorders) | 3
Posterior capsule opacification (Eye disorders) | 1
Presbyopia (Eye disorders) | 1
Pterygium (Eye disorders) | 1
Punctate keratitis (Eye disorders) | 1
Pupils unequal (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 3
Retinal vein occlusion (Eye disorders) | 1
Retinal vein thrombosis (Eye disorders) | 1
Scleral discolouration (Eye disorders) | 1
Scotoma (Eye disorders) | 1
Sicca syndrome (Eye disorders) | 37
Strabismus (Eye disorders) | 1
Trichiasis (Eye disorders) | 4
Vision blurred (Eye disorders) | 17
Visual impairment (Eye disorders) | 22
Vitreous haemorrhage (Eye disorders) | 1
Vitreous opacities (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 20
Dyspepsia (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 197
Tongue dry (Gastrointestinal disorders) | 1
Adverse drug reaction (General disorders) | 14
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Death (General disorders) | 3
Drug ineffective (General disorders) | 4
Drug intolerance (General disorders) | 5
Fatigue (General disorders) | 1510
Mucosal dryness (General disorders) | 1
Oedema peripheral (General disorders) | 1
Corneal graft rejection (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 873
Multiple allergies (Immune system disorders) | 1
Reaction to preservatives (Immune system disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Adenoviral conjunctivitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Chronic sinusitis (Infections and infestations) | 1
Herpes ophthalmic (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Corneal scar (Injury, poisoning and procedural complications) | 1
Blood pressure decreased (Investigations) | 4
Blood pressure increased (Investigations) | 2
Heart rate decreased (Investigations) | 1
Intraocular pressure decreased (Investigations) | 1
Intraocular pressure fluctuation (Investigations) | 2
Thyroid function test normal (Investigations) | 1
Weight decreased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2
Gout (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance disorder (Nervous system disorders) | 1
Cerebellar ischaemia (Nervous system disorders) | 1
Cerebrosclerosis (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 6
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 48
Dysgeusia (Nervous system disorders) | 17
Headache (Nervous system disorders) | 431
Memory impairment (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Parkinsonism (Nervous system disorders) | 1
Senile dementia (Nervous system disorders) | 1
Sensory disturbance (Nervous system disorders) | 1
Trigeminal neuralgia (Nervous system disorders) | 1
Affect lability (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 2
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 17
Emotional distress (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 2
Neurosis (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 8
Renal disorder (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 8
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 204
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 1
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 10
Ingrown hair (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 9
Yellow skin (Skin and subcutaneous tissue disorders) | 1
Treatment noncompliance (Social circumstances) | 22
Cardiac pacemaker insertion (Surgical and medical procedures) | 3
Cataract operation (Surgical and medical procedures) | 1
Corneal transplant (Surgical and medical procedures) | 1
Eye excision (Surgical and medical procedures) | 1
Eye laser surgery (Surgical and medical procedures) | 1
Eye operation (Surgical and medical procedures) | 1
Eye prosthesis insertion (Surgical and medical procedures) | 3
Intraocular lens implant (Surgical and medical procedures) | 1
Photocoagulation (Surgical and medical procedures) | 1
Angiosclerosis (Vascular disorders) | 1
Blood pressure inadequately controlled (Vascular disorders) | 2
Circulatory collapse (Vascular disorders) | 2
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 8
Peripheral coldness (Vascular disorders) | 2
Raynaud's phenomenon (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Except at baseline, number of subjects analyzed in treatment groups do not necessarily summarize to "All subjects" total; subjects drop out of treatment group when therapy changes. "All subjects" shows all subjects irrespective of any therapy change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.